CLINICAL TRIAL: NCT02310282
Title: Telemedicine for Optimized Collection of CLinical datA in Patients With Suspicion of Acute Stroke
Acronym: TeleCLASS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: B.U.N. 143201010021
Record Dates: First submitted 2014-12-01; First posted 2014-12-08 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2015-12

CONDITIONS: Stroke
Keywords: Telemedicine; Emergency medicine; Stroke; Stroke syndromes
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Telemedicine: In-hospital telemedicine by a stroke expert aiming to assess stroke severity using the Unassisted TeleStroke Scale.
  Interventions: Device: Telemedicine

INTERVENTIONS:
Device: Telemedicine — In-hospital telemedicine

SUMMARY:
Observational prospective single-center study on the discriminatory value of the Unassisted TeleStroke Scale for differentiation between patients with lacunar stroke and those with other acute stroke syndromes.

DETAILED DESCRIPTION:
Assessment of stroke severity and differentiation between large-artery and small-artery stroke is pivotal for adequate treatment decision taking. Patients with small vessel stroke tend have a better prognosis than those with large artery disease. Further, patients with small artery infarction (lacunar stroke) have shown to respond well to treatment with intravenous recombinant tissue plasminogen activator (IV rt-PA), but are poor candidates for endovascular recanalization. Conversely, IV rt-PA may be less effective at restoring perfusion of large artery occlusion, a stroke subtype that may benefit from intra-arterial thrombolysis or embolectomy. Similarly, patients with large intracerebral hemorrhage or cerebellar hemorrhage may require neurosurgical interventions, such as intracranial pressure monitoring, ventricular drainage, surgical evacuation, or hemicraniectomy.

The purpose of TeleCLASS is to evaluate the discriminatory value of the Unassisted TeleStroke Scale (UTSS) obtained through in-hospital telemedicine for differentiation between patients with lacunar stroke and those with other acute stroke syndromes (nonLACS).

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years
* Suspicion of acute stroke with symptom onset < 72 h before teleconsultation
* NIHSS score > 0
* Informed consent

Exclusion criterion:

* Patients for whom telestroke consultation would delay any diagnostic or therapeutic intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion of acute stroke admitted to the Emergency Department or the Stroke Unit of the Universitair Ziekenhuis Brussel
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Predictive validity of the UTSS for patient classification between lacunar syndromes and other stroke syndromes based on the Oxfordshire Community Stroke Project classification. | within 3 days
  Receiver operating curves, c-statistics, optimal thresholds, likelihood ratios and accuracy measures (sensitivity, specificity, positive predictive value, negative predictive value and overall accuracy) will be calculated to evaluate the predictive ability of the UTSS for discrimination between lacunar syndrome (LACS) and other stroke syndromes (nonLACS)

SECONDARY OUTCOMES:
Predictive validity of the UTSS for vessel status, classifying patients with acute ischemic stroke between those with large-artery occlusion and those without large-artery occlusion on imaging. | within 3 days
  Receiver operating curves, c-statistics, optimal thresholds, likelihood ratios and accuracy measures (sensitivity, specificity, positive predictive value, negative predictive value and overall accuracy) will be calculated to evaluate the predictive ability of the UTSS for discrimination between patients with large-artery occlusion and those without large-artery occlusion on imaging.
Predictive validity of the total UTSS score with cutoff value 6 for patient classification between lacunar syndromes and other stroke syndromes based on the Oxfordshire Community Stroke Project classification. | within 3 days
  Likelihood ratios and accuracy measures (sensitivity, specificity, positive predictive value, negative predictive value and overall accuracy) will be calculated to evaluate the predictive ability of the UTSS for discrimination between lacunar syndrome (LACS) and other stroke syndromes (nonLACS)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques De Keyser, MD PhD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Brussels Capital, Belgium